CLINICAL TRIAL: NCT06172335
Title: Effects of Ketolic Acid on Atherosclerosis Markers in High-risk Patients With Metabolic Syndrome (Effekt av Ketolinsyre på aterosklerosemarkører i høyrisikopasienter Med Metabolsk Syndrom)
Brief Title: Effects of Cetoleic Acid on Atherosclerosis (Ketolinsyre's Effekt på Aterosklerose)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Kirsten Bjørklund Holven, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 605236
Record Dates: First submitted 2023-10-02; First posted 2023-12-15 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Metabolic Syndrome
Keywords: Omega 3 fatty acids; Sustainability; Cetoleic acid; Very long monounsaturated fatty acid; Cardiovascular disease prevention; Antiinflammation
MeSH Terms: conditions — Metabolic Syndrome | interventions — cetoleic acid

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded controlled trial (Randomized 1:1, control:intervention).
  Run-in period of 3 weeks where all participants receive the control capsules.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All participant, the major investigator, study coordinator and the study staff are blinded for the randomizing. The capsules and capsule containers will only be identifiable by the ID (identifying) numbers on the containers.
  Allocation of participants to the specific intervention group is carried out by a statistician and one person not involved in conducting the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Cetoleic acid) (Experimental): 6 x capsules intervention oil (oil = mix of fish oils, olive oil, high-oleic sunflower oil and rapeseed oil) with high content of cetoleic acid (1780 mg/day, estimated: 29,76%) every morning for 4 weeks.
  Interventions: Dietary Supplement: Cetoleic acid
- Control oil (Placebo Comparator): 6 x capsules control oil (oil= mix of fish oils, olive oil, high-oleic sunflower oil and rapeseed oil) with low content of cetoleic acid (35 mg/day, estimated 0.58%) every morning for 4 weeks.
  Interventions: Dietary Supplement: Control oil

INTERVENTIONS:
Dietary Supplement: Cetoleic acid — Very long monounsaturated fatty acid (C22:1n-11)
  Arms: Intervention (Cetoleic acid)
Dietary Supplement: Control oil — Mix of oils with low cetoleic acid content
  Arms: Control oil

SUMMARY:
In this Randomized Controlled Trial (RCT) we want to study the effect of an oil with high concentrations of cetoelic acid (C22:n1-11) (intervention) compared to supplements with a low concentration of cetoleic acid (control), but with equivalent content of EPA og DHA, on plasma levels of epa and dha as well as atherosclerotic markers, glucose, c-peptide and triglycerides in a patient group with a metabolically unfavorable phenotype.

Our primary endpoints are changes in the concentration of EPA and DHA in plasma.

DETAILED DESCRIPTION:
This is a randomized double-blinded controlled trial (randomized 1:1). Study population: men and women 20-70 years with a metabolically unfavorable phenotype defined as: triglycerides > 1.7 mmol/L and waist measurement > 80 cm (women) and > 94 cm (men).

Study design:

* 3 weeks run-in-period where all participants consume control capsules every morning.
* Randomization intervention: control (1:1). All participants consume their capsules (control or intervention) for 4 weeks.

The intervention oil is consists of an oil high in cetoleic acid and the control oil is low in cetoleic acid. Both the intervention oil and the control oil are a mix of different oils; fish oils, olive oil, "high-oleic sunflower oil" and rapeseed oil so that the content of EPA, DHA and ALA is similar in the two oils.

Power calculation and sample size:

It was expected a difference of 15% in n-3 between the groups after the intervention (Østbye et al. 2019, doi:10.1017/S0007114519001478).

The level of significance was set to 5% (two-sided) and the power to 80%. A total of thirty-eight subjects were required to participate in the study, but a high dropout rate was expected (20%) and it was considered necessary to include a total of seventy (n=70) subjects (thirty-five per arm).

ELIGIBILITY:
Inclusion Criteria:

* Triglycerides > 1.7 mmol/L
* Waist measurement > 80 cm (women) and > 94 cm (men)

Exclusion Criteria:

* Chronic disease (liver/kidney/metabolism)
* Ongoing active cancer treatment
* Excessive alcohol consumption (>40g/day)
* Pregnant/breastfeeding or planned pregnancy during the intervention
* High intake of fish (>3 weekly meals)
* Level of free thyroxine (T4) and triiodothyronine (T3) outside reference ranges.
* Hypertension (≥ 160/ 100 mmHg)
* Total cholesterol > 7.8 mmol/L
* Blood donation during the intervention period
* Difficulty following the protocol
* Smoking or sniffing
* Regular use (> 1 day/week) of anti-inflammatory drugs
* Regular use of omega-3 supplements/cod liver oil
* Drug use other than stable use of statins, hypertension drugs (Ca antagonists, diuretics and beta blockers).
* Hormonal treatment excluding stable use of thyroxine and birth control pills/contraceptive rod

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
EPA and DHA in plasma | 4 weeks intervention
  EPA and DHA concentration in plasma measured at baseline and after 4 week intervention (and as a "control measurement" at the screening visit)

SECONDARY OUTCOMES:
Lipid profile | 4 weeks intervention
  Plasma levels of triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol, apolipoproteins (apoB and apoA), and Lp(a)
Glucose | 4 weeks intervention
  Serum levels of glucose
Inflammatory markers | 4 weeks intervention
  The concentration of circulating levels of inflammatory markers
Gene expression, metabolome and lipidome | 4 weeks intervention
  Changes in PBMC (peripheral blood mononuclear cell) gene expression profile. Changes in plasma metabolome and lipidome profile. Changes in PBMC epitranscriptome, as a regulator of the gene expression profile
Resolvin | 4 weeks intervention
  Blood levels of resolvin (omega- 3 derivates) concentration
C-peptid | 4 weeks intervention
  serum levels of C-peptid

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten B. Holven, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway